CLINICAL TRIAL: NCT07364279
Title: Effect of Wii Fit Balance Board Games on Balance in Patients With Osteoporosis Post Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, linda raafat daniel, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/003323; Linda Raafat Daniel (Registry Identifier: Linda Raafat Daniel)
Record Dates: First submitted 2025-06-10; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Osteoporosis; Mastectomy
Keywords: osteoporosis post mastectomy; females; balance; EFFECT OF WII FIT BALANCE BOARD GAMES
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Wii Fit group (Experimental): This group includes thirty female patients suffering from balance dysfunction resulting from osteoporosis post mastectomy. They will receive Wii Fit balance board exercises for 3 sessions per week for 8 weeks, in addition to traditional balance exercises and the routine medical treatment.
  Interventions: Device: Wii fit balance board; Other: traditional balance exercise; Drug: Calcium supplement
- Control group: (Active Comparator): This group includes thirty female patients suffering from balance dysfunction resulting from osteoporosis post mastectomy. They will receive traditional balance exercises in addition to the routine medical treatment for 3 sessions per week for 8 weeks.
  Interventions: Other: traditional balance exercise; Drug: Calcium supplement

INTERVENTIONS:
Device: Wii fit balance board — Wii fit balance board Compose of Hardware which comprised of a regular PC, a 10" LCD screen and a Wii Fit balance board. The correspondence between this device and the screen was set up by means of Bluetooth convention. Along these lines, the activities run on a PC and the framework utilized the WBB as interface. A platform has sensors that action weight and center point of gravity . The software is Darwiin Remote . The average displacement of the center of gravity was determined to assess the equilibrium status. The force plate has 4 strain gauges and can measure the tension got from changes in posture and was associated with a PC screen. The center of gravity point can be shown on the screen to give a client visual input and to gauge the equilibrium status. The four sensors yet to be determined board can detect weight changes and show the distribution of body weight. The 4 sensors measure weightcan be added to get the body loads of individual clients.
  Arms: Study group (Wii Fit group
Other: traditional balance exercise — traditional balance exercise
Drug: Calcium supplement — traditional treatment
  Other Names: vitamens

SUMMARY:
This study will be a randomized controlled trial. The purpose of the study is to evaluate the therapeutic effect of Wii Fit balance board games on balance in patients with osteoporosis post mastectomy.

DETAILED DESCRIPTION:
Women with breast cancer face an increased risk of osteoporosis, necessitating screening and treatment to prevent fractures due to aging and treatment effects. Osteoporosis exacerbates balance issues, raising fall risks among these patients. The treatments often lead to accelerated bone loss and compromised musculoskeletal support, amplifying their vulnerability to fractures. Integrated management strategies that enhance bone health and balance rehabilitation are essential for this group. Post-mastectomy systematic movement exercises are vital for maintaining activity and preventing posture issues, significantly improving balance. Additionally, the use of interactive systems like Wii Fit has shown to effectively aid balance training and improve overall physical function for breast cancer patients, making it a valuable component of at-home rehabilitation programs to reduce fall risk and enhance quality of life.

ELIGIBILITY:
Inclusion Criteria:

* The subject selection will be according to the following criteria:

  1. All patients are female.
  2. Age ranges from 40_60 years.
  3. All patients suffering from balance dysfunctions resulting from osteoporosis after mastectomy.
  4. All participants will have informed consent to participate in this study.
  5. All patients will participate in the study after 6 months of receiving chemotherapy and diagnosed with osteoporosis.
  6. All patients will follow the same diet .
  7. Ability to stand and ambulate independently

Exclusion Criteria:

* Patients will be excluded from the study if they met any of the following criteria:

  1. Patients with visual or hearing, vestibular impairment. 25
  2. Patients with Previous breast cancer surgery on the present or contralateral side.
  3. Patients receiving hormonal therapy
  4. Patients with Active or metastatic cancer focus.
  5. Patients with Venous thrombosis.
  6. Osteoarticular and/or Rheumatological disorders, significantly disturbing balance.
  7. Patients with severe orthopedic injuries to the lower extremities (e.g. Ankle fracture, joint fusion or joint replacement).
  8. Patients with neurological disturbances that cause impaired balance such as hemiparesis, ataxia, vertigo and vestibular disturbances.
  9. Patients with mental disorders.
  10. Pregnant patients.
  11. Patients with diabetes mellitus.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-11-05 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale (BBS). | at baseline and after 8 weeks
  The Berg Balance Scale consists of 14 items, each scored on an ordinal scale from 0 to 4 (0 = unable to perform, 4 = normal performance). Document the baseline scores for each item.
  Tasks Included:
  Sitting balance. Standing balance. Dynamic balance.
  Scoring:
  Total possible score is 56 points. Higher scores indicate better balance.
  Post-Treatment Assessment:
  Re-evaluate the patient using the same BBS after eight weeks of treatment.

SECONDARY OUTCOMES:
assessment of balance using the Wii Fit balance board | at baseline and after 8 weeks
  Instruct the patient to stand on the Wii Fit balance board. Measure the center of pressure (COP) results.
  The balance board estimates the pressure contributed by the left and right halves of the body. Ideal center of pressure proportion is 50/50 or 1.00 Instruct the patient to stand on the Wii Fit balance board.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arshad, H., Khattak, H., Anwar, K., Majeed, Y., & Malakandi, H. B. (2022). Comparison of exergames versus traditional balance exercise to improve balance and reduce risk of falls in chronic stroke patients. Journal of Medical Sciences (Peshawar), 30, 134- 138. https://doi.org/10.52764/jms.22.30.2.7 Blackie, R. (2020). Diagnosis, assessment and management of osteoporosis. Prescriber, 31, 14-19. https://doi.org/10.1002/psb.1815 Cabanas-Valdés, R., Boix-Sala, L., Grau-Pellicer, M., Guzmán-Bernal, J. A., Caballero-Gómez, F. M., & Urrútia, G. (2021). The Effectiveness of Additional Core Stability Exercises in Improving Dynamic Sitting Balance, Gait and Functional Rehabilitation for Subacute Stroke Patients (CORE-Trial): Study Protocol for a Randomized Controlled Trial. International Journal of Environmental Research and Public Health, 18(12), 6615. https://doi.org/10.3390/ijerph18126615 Castañeda, S., Casas, A., González-del-Alba, A., Martínez-Díaz-Guerra, G., Nogués, X., Ojeda Thies, C., Torregrosa Suau, Ó., & Rodríguez-Lescure, Á. (2022). Bone loss induced by cancer treatments in breast and prostate cancer patients. Clinical & 37 Translational Oncology, 24(11), 2090-2106. https://doi.org/10.1007/s12094-022-02872-1 Choksi, P., Williams, M., Clark, P. M., & Van Poznak, C. (2013). Skeletal Manifestations of Treatment of Breast Cancer. Current Osteoporosis Reports, 11(4), 319-328. https://doi.org/10.1007/s11914-013-0179-7 Clynes, M. A., Cooper, C., Dennison, E. M., Jacobsen, B. K., & Javaid, M. K. (2020). The epidemiology of osteoporosis. British Medical Bulletin, 133(1), 105-117. Czajka, M. L., & Pfeifer, C. (2024). Breast Cancer Surgery. In StatPearls. StatPearls Publishing. http://www.ncbi.nlm.nih.gov/books/NBK553076/ Deans, S. M. (2011). Determining the validity of the Nintendo Wii balance board as an assessment tool for balance. https://doi.org/10.34917/2820752 Doruk Analan, P., & Kaya, E. (2019). Postural Stability in Patients with Lower Li